CLINICAL TRIAL: NCT04835610
Title: The Comparison of the Effectiveness of Finger and Forehead Plethysmographic Variability Index Monitoring in Pediatric Patients
Brief Title: Effectiveness of Finger and Forehead Plethysmographic Variability Index Monitoring in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Other Study IDs: 09.2020.132
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: PVI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- PVI values: PVI values measured at the finger and forehead areas in pediatric patients
  Interventions: Device: pvi
- no control group: no control group
  Interventions: Device: pvi

INTERVENTIONS:
Device: pvi — The Plethysmographic Variability Index (PVI) can be measured with both finger and forehead probes. Vasoconstriction may reduce the reliability of PVI measurements in pediatric surgical patients prone to hypothermia. The vascular structure of the forehead area is resistant to changes in vasomotor tonus. The aim of our study is to compare the efficacy of PVI values measured at the finger and forehead areas to predict fluid responsiveness in these patients.

SUMMARY:
In pediatric surgical patients, the sensitivity of forehead and finger PVI monitoring was similar for the prediction of fluid responsiveness, whereas the specificity of forehead monitoring was higher. The use of forehead PVI probes in the fluid management of these patients seemed to be appropriate because cephalic region was not affected by low perfusion states.

DETAILED DESCRIPTION:
he Plethysmographic Variability Index (PVI) can be measured with both finger and forehead probes. Vasoconstriction may reduce the reliability of PVI measurements in pediatric surgical patients prone to hypothermia. The vascular structure of the forehead area is resistant to changes in vasomotor tonus. The aim of our study is to compare the efficacy of PVI values measured at the finger and forehead areas to predict fluid responsiveness in these patients.

Fifty pediatric patients with obtained parental consent and ethics committee approval underwent elective minor surgery were included into the study. Basic monitoring, finger and forehead perfusion index (PI) and PVI monitoring were applied. Hemodynamic parameters, PI, PVI, cardiac output (CO) values were recorded. The 15% increase in CO with passive leg raise (PLR) maneuver was estimated as fluid responsiveness. Two groups were created: Group R (fluid responsive); Group NR (fluid nonresponsive). Mann-Whitney U, t, chi-square and ROC tests were used in statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

written consent from their parents patients undergoing elective minor surgery with bleeding less than 500ml Children between the ages of 5-12.

Exclusion Criteria:

those who stay in the specified age range those with cardiopulmonary disease spontaneous breathing positive allen test peripheral circulatory failure vasopressor therapy anemia hypothermic

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: pediatric patients
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
The Plethysmographic Variability Index (PVI) | 15 minute intervals during surgery
  The Plethysmographic Variability Index (PVI) can be measured with both finger and forehead probes by pvi monitoring.

SECONDARY OUTCOMES:
Cardiac output (CO) | 15 minute intervals during surgery
  Cardiac output (CO) values were recorded by noninvasive cardiac output monitoring

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided